CLINICAL TRIAL: NCT04539223
Title: Study of Lipids Inside the Carotid With Evolocumab: A Randomized Trial of Evolocumab on Carotid Artery Atherosclerotic Plaque Morphology Prior to Carotid EndArterectomy (SLICE-CEA CardioLink-8 Study)
Brief Title: A Study of Evolocumab on Carotid Artery Atherosclerotic Plaque Morphology Prior to Carotid EndArterectomy
Acronym: SLICE-CEA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Canadian Medical and Surgical Knowledge Translation Research Group (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLICE-CEA-001
Record Dates: First submitted 2020-08-30; First posted 2020-09-04 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Carotid Artery Stenosis; Asymptomatic Carotid Artery Stenosis
Keywords: CEA; Carotid EndArterectomy; Evolocumab; Carotid Artery
MeSH Terms: conditions — Carotid Stenosis | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: Twenty-six week treatment with or without evolocumab in addition to current medical management.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug (Evolocumab) (Active Comparator): Individuals randomized to this arm will administer Evolocumab subcutaneously (SC) every two weeks (Q2W) for 26 weeks.
  Interventions: Drug: Evolocumab
- No Drug (Standard of Care) (No Intervention): Individuals randomized to this arm will not administer a placebo.

INTERVENTIONS:
Drug: Evolocumab — Autoinjector 1-mL deliverable volume of 140 mg/mL
  Arms: Drug (Evolocumab)

SUMMARY:
This is a multicenter, randomized, open label study with blinded outcome assessment to evaluate the impact of additional/intensive LDL-cholesterol reduction with evolocumab on carotid artery atherosclerotic plaques in higher risk subjects with severe asymptomatic but vulnerable plaques.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years old
2. Significant (70-99%) carotid artery stenosis on one side, as measured by duplex ultrasound or angiogram
3. Asymptomatic carotid stenosis (no history of ipsilateral stroke or TIA within 180 days)
4. Deemed to be fit for carotid endarterectomy
5. At least one of the following high-risk features: (a) prior stroke >6months prior to randomization; (b) peripheral artery disease; (c) current smoker; (d) type 2 diabetes; (e) eGFR ≥ 30 mL/min/1.73m2 and <60 ml/min/1.73m2; (f) hsCRP > 2mg/L in the absence of alternative known causes of hsCRP elevations including autoimmune diseases or active infections.
6. On a moderate to high intensity statin therapy (defined as atorvastatin 40-80mg daily, rosuvastatin 20-40mg or simvastatin 40mg daily) unless a lower dose, or another statin or non-statin therapy is clinically justified

Exclusion Criteria:

1. Contraindications for MRI (pacemaker; neurostimulator; non-removable metal fragments in the eye; etc.)
2. Patients in whom additional lowering of LDL-C with evolocumab is deemed to be clinically inappropriate
3. Currently taking simvastatin >40mg/day
4. High risk comorbidities such as severe heart failure, severe COPD, severe renal disease, known severe hepatic impairment, unstable coronary syndrome, and/or advanced dementia
5. eGFR <30 mL/min/1.73m2
6. Current, prior within past year, or known planned use of PCSK9 inhibition treatment
7. Known intolerance or allergy to evolocumab or other PCSK9 inhibitors
8. Known latex allergy
9. Women who are pregnant or breastfeeding
10. Women of child bearing potential who are unwilling to use proper family planning or birth control methods to avoid pregnancy. Women are considered post-menopausal and not of childbearing potential after 12 months of natural (spontaneous) amenorrhea or have had a surgical procedure such as hysterectomy which makes pregnancy impossible
11. Inability to comply with protocol-required study visits or procedures, including administration of study drug
12. Severe concomitant disease that is expected to reduce life expectancy to less than 5 years
13. Participation in another investigational device or drug study which is likely to affect the primary outcome, within 30 days of planned initiation of study drug

Additional Inclusion Criteria

If all eligibility criteria listed above are met, participants with only one high risk feature will undergo a time-of-flight MR angiogram, where one additional inclusion criteria will be assessed to confirm eligibility:

1. Evidence of IPH on MRI

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Change in lipid rich necrotic core (LRNC) volume | Baseline to end of treatment (average of 6 months)
  As measured by MRI

SECONDARY OUTCOMES:
Change in vessel wall volume | Baseline to end of treatment (average of 6 months)
  As measured by MRI
Change in vessel lumen volume | Baseline to end of treatment (average of 6 months)
  As measured by MRI

OTHER OUTCOMES:
Plaque Histology and Morphology | At the end of treatment (average of 6 months)
  Obtained at time of CEA
Lipid Levels | Baseline to end of treatment (average of 6 months)
  Serum lipid levels

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Al-Omran, MD, Principal Investigator — Unity Health Toronto
Locations (3):
- Canada (3):
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - East Toronto Vascular Clinic, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario